CLINICAL TRIAL: NCT07020533
Title: A Phase 1b Trial of CMV-MVA Triplex Vaccine in Haploidentical Stem Cell Donors and Recipients to Enhance CMV-Specific Immunity and Prevent CMV Viremia in Recipients of Hematopoietic Stem Cell Transplant
Brief Title: A Vaccine (CMV-MVA Triplex Vaccine) for the Enhancement of CMV-Specific Immunity and the Prevention of CMV Viremia in Patients Undergoing Haploidentical Hematopoietic Stem Cell Transplant
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 24168; NCI-2025-03633 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24168 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-06-06; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Accelerated Phase Chronic Myeloid Leukemia, BCR-ABL1 Positive; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Lymphocytic Leukemia; Chronic Phase Chronic Myeloid Leukemia, BCR-ABL1 Positive; Hematopoietic and Lymphatic System Neoplasm; Hodgkin Lymphoma; Lymphoblastic Lymphoma; Myelodysplastic Syndrome; Myelofibrosis; Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Hodgkin Disease; Myelodysplastic Syndromes; Primary Myelofibrosis; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin | interventions — Specimen Handling; Stem Cell Transplantation; letermovir; Bone Marrow Purging; Blood Component Removal; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Donors (CMV-MVA Triplex vaccine, G-CSF) (Experimental): Participants receive CMV-MVA Triplex vaccine IM once and then receive G-CSF on study. Additionally, participants undergo apheresis on study as well as blood sample collection on study and may optionally undergo blood sample collection during follow up.
  Interventions: Procedure: Biospecimen Collection; Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine; Procedure: Pheresis; Biological: Recombinant Granulocyte Colony-Stimulating Factor
- Recipients, Modality 1 (CMV-MVA Triplex vaccine, letermovir) (Experimental): Patients receive myeloablative conditioning during screening and undergo HCT from haploidentical vaccinated donor on day 0. Patients receive CMV-MVA Triplex vaccine IM QD on days 28, 56 and 100 and receive letermovir IV over 1 hour or PO QD on days 7 to 100. Treatment continues in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Procedure: Haploidentical Hematopoietic Cell Transplantation; Drug: Letermovir; Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine; Procedure: Myeloablative Conditioning
- Recipients, Modality 2 (CMV-MVA Triplex vaccine, letermovir) (Experimental): Patients receive myeloablative conditioning during screening and undergo HCT from haploidentical vaccinated donor on day 0. Patients receive CMV-MVA Triplex vaccine IM QD on days 28, 56 and 100 and receive letermovir IV over 1 hour or PO QD on days 7 to 28. Treatment continues in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Procedure: Haploidentical Hematopoietic Cell Transplantation; Drug: Letermovir; Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine; Procedure: Myeloablative Conditioning
- Recipients, Modality 3 (CMV-MVA Triplex vaccine) (Experimental): Patients receive myeloablative conditioning during screening and undergo HCT from haploidentical vaccinated donor on day 0. Patients receive CMV-MVA Triplex vaccine IM QD on days 28, 56 and 100. Treatment continues in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Procedure: Haploidentical Hematopoietic Cell Transplantation; Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine; Procedure: Myeloablative Conditioning

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Ancillary studies
  Arms: Recipients, Modality 1 (CMV-MVA Triplex vaccine, letermovir); Recipients, Modality 2 (CMV-MVA Triplex vaccine, letermovir); Recipients, Modality 3 (CMV-MVA Triplex vaccine)
Procedure: Haploidentical Hematopoietic Cell Transplantation — Undergo HCT
  Other Names: Haploidentical Stem Cell Transplantation; HLA-Haploidentical Hematopoietic Cell Transplantation; Stem Cell Transplantation, Haploidentical
  Arms: Recipients, Modality 1 (CMV-MVA Triplex vaccine, letermovir); Recipients, Modality 2 (CMV-MVA Triplex vaccine, letermovir); Recipients, Modality 3 (CMV-MVA Triplex vaccine)
Drug: Letermovir — Given IV or PO
  Other Names: 2-((4S)-8-Fluoro-2-(4-(3-methoxyphenyl)piperazin-1-yl)-3-(2-methoxy-5-(trifluoromethyl)phenyl)-4H-quinazolin-4-yl)acetic Acid; AIC246; MK-8228; Prevymis
  Arms: Recipients, Modality 1 (CMV-MVA Triplex vaccine, letermovir); Recipients, Modality 2 (CMV-MVA Triplex vaccine, letermovir)
Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine — Given IM
  Other Names: CMV-MVA Triplex Vaccine; Multi-antigen CMV-Modified Vaccinia Ankara Vaccine
Procedure: Myeloablative Conditioning — Receive myeloablative conditioning
  Other Names: Myeloablation; Myeloablative; Myeloablative Cytoreduction
  Arms: Recipients, Modality 1 (CMV-MVA Triplex vaccine, letermovir); Recipients, Modality 2 (CMV-MVA Triplex vaccine, letermovir); Recipients, Modality 3 (CMV-MVA Triplex vaccine)
Procedure: Pheresis — Undergo apheresis
  Other Names: Apheresed; Apheresis; Blood Component Removal; Collection, Apheresis/Leukapheresis; Hemapheresis
  Arms: Donors (CMV-MVA Triplex vaccine, G-CSF)
Biological: Recombinant Granulocyte Colony-Stimulating Factor — Given G-CSF
  Other Names: Recombinant Colony-Stimulating Factor 3; rhG-CSF
  Arms: Donors (CMV-MVA Triplex vaccine, G-CSF)

SUMMARY:
This phase Ib trial tests the safety, side effects, and how well cytomegalovirus (CMV)-modified vaccinia Ankara (MVA) Triplex vaccine works in enhancing CMV-specific immunity and preventing CMV viremia in patients undergoing haploidentical hematopoietic stem cell transplant. Haploidentical stem cell transplantation (haploHCT) has advanced to become the predominant procedure for patients lacking a matched donor. Compared to matched related donor transplants, the rate of significant CMV infection is higher in patients undergoing a haploHCT. Significant CMV infection is associated with an increased risk of complications and death. Vaccination is the main preventative approach to limit complications and death in immunocompromised patients at high risk of post-stem cell transplant infections. CMV-MVA Triplex vaccine, is a CMV vaccine based on the attenuated poxvirus, modified vaccinia Ankara (MVA), developed to enhance CMV-specific immunity in both healthy stem cell transplant donors and stem cell transplant patients to prevent significant CMV infection post-stem cell transplant. Giving CMV-MVA triplex vaccine may be safe, tolerable and/or effective in enhancing cytomegalovirus (CMV)-specific immunity and preventing CMV viremia in patients undergoing a haploHCT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether the multi-peptide cytomegalovirus-modified vaccinia Ankara vaccine (CMV-MVA Triplex [Triplex]) vaccination of stem cell donors (D) and recipients (R) alone or in combination with letermovir safely protects against CMV events for day (d)100 in the absence of preemptive therapy (PET) and to determine the recommended duration of letermovir use as phase 2 modality in the haploidentical stem cell transplantation (haploHCT)-R.

SECONDARY OBJECTIVES:

I. To evaluate safety of Triplex in the haploHCT-R. II. To evaluate cumulative incidence of CMV events up to d180 post-hematopoietic stem cell transplant (HCT).

III. To evaluate CMV viremia levels over time in the HCT-R. IV. To evaluate cumulative incidence of CMV disease. V. To evaluate use of PET by the HCT-R.

EXPLORATORY OBJECTIVES:

I. To assess levels and durability of CMV specific T cell immunity. II. To assess polyfunctional T cell responses and cell-surface memory markers until d180 post-HCT.

OUTLINE:

DONORS: Participants receive CMV-MVA Triplex vaccine intramuscularly (IM) once and then receive granulocyte colony stimulating factor (G-CSF) on study. Additionally, participants undergo apheresis on study as well as blood sample collection on study and may optionally undergo blood sample collection during follow up.

RECIPIENTS: Patients are assigned to 1 of 3 modalities.

MODALITY 1: Patients receive myeloablative conditioning during screening and undergo HCT from haploidentical vaccinated donor on day 0. Patients receive CMV-MVA Triplex vaccine IM once daily (QD) on days 28, 56 and 100 and receive letermovir intravenously (IV) over 1 hour or orally (PO) QD on days 7 to 100. Treatment continues in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the study.

MODALITY 2: Patients receive myeloablative conditioning during screening and undergo HCT from haploidentical vaccinated donor on day 0. Patients receive CMV-MVA Triplex vaccine IM QD on days 28, 56 and 100 and receive letermovir IV over 1 hour or PO QD on days 7 to 28. Treatment continues in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the study.

MODALITY 3: Patients receive myeloablative conditioning during screening and undergo HCT from haploidentical vaccinated donor on day 0. Patients receive CMV-MVA Triplex vaccine IM QD on days 28, 56 and 100. Treatment continues in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 2 weeks until day 180 and then at day 365.

ELIGIBILITY:
Inclusion Criteria:

* DONORS: Documented informed consent of the participant. This can be done in person or informed consent can be obtained remotely.

  * Remote consent, when appropriate, will be obtained per institutional guidelines.
  * Assent, when appropriate, will be obtained per institutional guidelines.
  * Adult subjects who require a legally authorized representative (LAR) will not be permitted to be enrolled under this protocol.
* DONORS: Age: 18 - 75.
* DONORS: Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* DONORS: Agreement by females and males of childbearing potential* to use an effective method of birth control (hormonal or barrier method) or abstain from heterosexual activity prior to study entry and for up to 90 days post-vaccination.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).
* RECIPIENTS: Documented informed consent of the participant and/or legally authorized representative. This can be done in person or informed consent can be obtained remotely.

  * Remote consent, when appropriate, will be obtained per institutional guidelines.
  * Assent, when appropriate, will be obtained per institutional guidelines.
  * Adult subjects who require a legally authorized representative (LAR) will not be permitted to be enrolled under this protocol.
* RECIPIENTS: Participant must be willing to comply with study and/or follow-up procedures, including willingness to be followed for one year post-HCT.
* RECIPIENTS: Age: 18 - 75.
* RECIPIENTS: Planned peripheral blood stem cell (PBSC) or bone marrow (BM) HCT for the treatment of the following hematologic malignancies:

  * Lymphoma (Hodgkin and Non-Hodgkin).
  * Myelodysplastic syndrome.
  * Acute lymphoblastic leukemia in first or second remission (for acute lymphoblastic leukemia/lymphoblastic lymphoma, the disease status must be in hematologic remission by bone marrow and peripheral blood. Persistent lymphadenopathy on computed tomography (CT) or CT/positron emission tomography(PET) scan without progression is allowed.)
  * Acute myeloid leukemia in first or second remission.
  * Chronic myelogenous leukemia in first chronic or accelerated phase, or in second chronic phase.
  * Other hematologic malignancies judged appropriate by the clinical principal investigators (PIs), including chronic lymphocytic leukemia, myeloproliferative disorders and myelofibrosis. Patients with multiple myeloma and those with non-malignant disease such as aplastic anemia are excluded**.

    * Adult cases of multiple myeloma (MM) are excluded as HCT is not standard of care for MM and is only performed in very advanced cases with an associated high risk of relapse and non-relapse mortality (NRM). Adults with aplastic anemia are excluded because their standard management includes T cell depletion with agents such as antithymocyte globulin (ATG), which is not permissible on this protocol. Patients undergoing a second haploHCT are not eligible (patients who have undergone a previous autologous HCT are eligible).
* RECIPIENTS: Patients receiving myeloablative (MA) or reduced intensity conditioning (RIC) are allowed.
* RECIPIENTS: CMV seropositive.
* RECIPIENTS: Eligible haploidentical donors will have 2-4 mismatches if human leukocyte antigen (HLA)-A, -B, -C, and -DRB1 typing is used; 2-5 mismatches if HLA-A, -B, -C, -DRB1, and -DQB1 typing is used; and 2-6 mismatches if HLA-A, -B, -C, -DRB1, -DQB1, and -DPB1 typing is used. A unidirectional mismatch in either the graft versus host or host versus graft direction is considered a mismatch. The donor and recipient must demonstrate that they are a full haplotype match by being identical at a minimum of one allele (at high resolution deoxyribonucleic acid [DNA]-based typing) at the following genetic loci: HLA-A, -B, -C, and DRB1 if 8 allele typing is used; HLA-A, -B, -C, -DRB1, and -DQB1 if 10 allele typing is used; and HLA-A, -B, -C, -DRB1-, DQB1, and -DPB1 is 12 allele typing is used.
* RECIPIENTS: Planned HCT with minimal to no-T cell depletion of graft.
* RECIPIENTS: Conditioning and immunosuppressive regimens according to institutional guidelines are permitted.
* RECIPIENTS: Total bilirubin ≤ 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease) (to be performed within 45 days prior to day 1 of protocol therapy).
* RECIPIENTS: Aspartate aminotransferase (AST) =< 2.5 x ULN (to be performed within 45 days prior to day 1 of protocol therapy).
* RECIPIENTS: Alanine aminotransferase (ALT) =< 2.5 x ULN (to be performed within 45 days prior to day 1 of protocol therapy).
* RECIPIENTS: Estimated creatinine clearance acceptable per institutional guidelines (to be performed within 45 days prior to day 1 of protocol therapy).
* RECIPIENTS: Left ventricular ejection fraction (LVEF) ≥ 50%.

  * Note: To be performed within 45 days prior to day 1 of protocol therapy.
* RECIPIENTS: If able to perform pulmonary function tests: forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and carbon monoxide diffusing capability (DLCO) (diffusion capacity) ≥ 50% of predicted (corrected for hemoglobin).

  * If unable to perform pulmonary function tests: Oxygen (O2) saturation > 92% on room air.
  * Note to be performed within 45 days prior to day 1 of protocol therapy.
* RECIPIENTS: Seronegative for HIV antigen (Ag)/antibody (Ab) combination (combo), hepatitis c virus (HCV)*, active hepatitis b virus (HBV) (surface antigen negative) and syphilis (RPR) within 2 months of registration and no history of disseminated cutaneous human papillomavirus (HPV) related disease.

  * If seropositive for HIV, HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetectable.
* RECIPIENTS: Meets other institutional and federal requirements for infectious disease titer requirements.

  * Note Infectious disease testing to be performed within 45 days prior to day 1 of protocol therapy.
* RECIPIENTS: Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (to be performed within 45 days prior to day 1 of protocol therapy).
* RECIPIENTS: Agreement by females and males of childbearing potential* to use an effective method of birth control (hormonal or barrier method) or abstain from heterosexual activity prior to study entry and up to 90 days post-HCT.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).

Exclusion Criteria:

* DONORS: Any prior transplant to day 1 of protocol therapy (day 1 defined as the day after donors receive the Triplex vaccine).
* DONORS: Chemotherapy, radiation therapy, biological therapy, immunotherapy within 21 days prior to day 1 of protocol therapy.
* DONORS: Receipt of any vaccine (licensed or investigational) within 30 days prior to and after the study vaccine.
* DONORS: Unfit to undergo standard stem cell mobilization and apheresis e.g. abnormal blood counts, history of stroke, uncontrolled hypertension.
* DONORS: Sickling hemoglobinopathy including hemoglobin (Hb)SS, HbAS, HbSC.
* DONORS: Donors with impaired cardiac function are excluded. Electrocardiography is routine for potential HCT donors over 60 years old and those with a history of heart disease. Subjects in whom cardiac function is abnormal (excluding 1st degree branch block, sinus bradycardia, sinus tachycardia or non-specific T wave changes) are ineligible for Triplex vaccination.
* DONORS: Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the donation procedure unlikely and making informed consent impossible.
* DONORS: Females only: Pregnant or breastfeeding.
* DONORS: Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* DONORS: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).
* RECIPIENTS: Any prior investigational CMV vaccine.
* RECIPIENTS: Experimental anti-CMV chemotherapy in the last 6 months.
* RECIPIENTS: Live attenuated vaccines (planned medications from the time of HCT to day 70 post-HCT).
* RECIPIENTS: Medically indicated subunit (Engerix-B for HBV; Gardasil for HPV) or killed vaccines (e.g. influenza, pneumococcal, or allergy treatment with antigen injections) (planned medications from the time of HCT to day 70 post-HCT).
* RECIPIENTS: Allergy treatment with antigen injections (planned medications from the time of HCT to day 70 post-HCT).
* RECIPIENTS: Alemtuzumab or any equivalent in vivo T-cell depleting agent (or CD34+ selection) (planned medications from the time of HCT to day 70 post-HCT).
* RECIPIENTS: Antiviral medications with known therapeutic effects on CMV such as ganciclovir (GCV)/valganciclovir (VAL), foscarnet (FOS), cidofovir, CMX-001, maribavir. Acyclovir has no known therapeutic efficacy against CMV and is allowable as standard of care to prevent herpes simplex virus (HSV) (planned medications from the time of HCT to day 70 post-HCT).
* RECIPIENTS: Prophylactic therapy with CMV immunoglobulin or prophylactic antiviral CMV treatment EXCEPT letermovir prophylaxis (prior to day 100) (planned medications from the time of HCT to day 70 post-HCT).
* RECIPIENTS: Disease-based radiation therapy (not total body irradiation) (planned medications from the time of HCT to day 70 post-HCT).
* RECIPIENTS: Other investigational product(s) - concurrent enrollment in other clinical trials using any investigational new drug (IND) drugs with unknown effects on CMV or with unknown toxicity profiles is prohibited (planned medications from the time of HCT to day 70 post-HCT).
* RECIPIENTS: Other medications that might interfere with the evaluation of the investigational product (planned medications from the time of HCT to day 70 post-HCT).
* RECIPIENTS: Patients with active autoimmune conditions requiring systemic immunosuppressive therapy within the previous 5 years.
* RECIPIENTS: Patients considered by PI/consenting physicians to have a complicated prior therapy or HCT regimen, or who have a low survival probability (e.g., refractory leukemia and/or undergoing 2nd HCT).
* RECIPIENTS: Poor risk disease/disease status including: Chronic myelogenous leukemia (CML) in blast crisis, acute myeloid leukemia (AML)/acute lymphoblastic leukemia (ALL) beyond 2nd remission, multiple myeloma, and aplastic anemia.
* RECIPIENTS: Females only: Pregnant or breastfeeding.
* RECIPIENTS: Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* RECIPIENTS: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-05-08 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Cytomegalovirus (CMV) reactivation prompting antiviral therapy | From day 0 to day 100 post-hematopoietic stem cell transplant (HCT)
  Will evaluate for CMV reactivation prompting antiviral therapy. Will be evaluated in patients that received a stem cell infusion from a Triplex vaccinated haploidentical donor and received the first Triplex vaccination.
CMV disease | From day 0 to day 100 post-HCT
  Will evaluate for CMV disease based on histology. Will be evaluated in patients that received a stem cell infusion from a Triplex vaccinated haploidentical donor and received the first Triplex vaccination.

SECONDARY OUTCOMES:
Unacceptable toxicity | Up to 28 days after the last Triplex vaccination
  Will evaluate for grade 3-4 adverse events based on Common Terminology Criteria for Adverse Events version 5.0 probably or definitely attributable to vaccination in both recipients and donors. Descriptive statistics will be used to summarize recipients and donor adverse events.
Serious adverse events (SAE) | Up to 365 days after Triplex vaccination
  Will evaluate for SAEs that are at least possibly related to Triplex vaccination in donors.
Incidence of acute graft-versus-host disease (GVHD) | Up to day 180 post-HCT
  Will evaluate for grade 3-4 acute GVHD. Documented/biopsy proven acute GVHD is graded according to Mount Sinai Acute GVHD International Consortium (MAGIC) grading. Cumulative incidence curves will be used to estimate acute GVHD.
Non-relapse mortality (NRM) | From HCT to death from other causes than disease relapse or progression, assessed up to day 180 post-HCT
  Will evaluate occurrence of NRM. Cumulative incidence curves will be used to estimate NRM.
CMV events | Up to day 180 post-HCT
  Will evaluate for CMV events. Death or relapse/progression prior to day 180 post-HCT will be counted as competing risk events. Patients who are alive and free of CMV events and relapse/progression at the last follow-up or day 180 post-HCT, whichever comes first, will be censored. Cumulative incidence curves will be used to estimate CMV events.
CMV viremia | From HCT to the date of two consecutive CMV quantitative polymerase chain reaction (qPCR) > 500 gc/mL/465 IU/mL, single event of CMV qPCR > 1500 CMV gc/mL/1,395 IU/mL, or CMV disease, whichever occurs first, assessed up to day 180 post-HCT
  Will evaluate for CMV viremia. Cumulative incidence curves will be used to estimate CMV viremia.
Incidence of late CMV viremia | From HCT to the date of two consecutive CMV qPCR > 500 gc/mL/465 IU/mL, single event of CMV qPCR > 1500 CMV gc/mL/1,395 IU/mL, or CMV disease, whichever occurs first, assessed from day 100 to day 365 post-HCT
  Will evaluate for incidence of late CMV viremia. Cumulative incidence curves will be used to estimate CMV viremia.
Neutrophil engraftment | From HCT to the first of 3 consecutive days with neutrophil count ≥ 0.5 X 10^3/uL
  Will evaluate time to neutrophil engraftment.
Platelet engraftment | From HCT to the first day of platelet count ≥ 20 X 10^3/uL independent of platelet transfusion support (date should reflect no transfusions in previous 7 days, and the first of 3 consecutive lab values on different days)
  Will evaluate time to platelet engraftment.
Incidence of severe acute GVHD | Up to day 180 post-HCT
  Will evaluate for grade 2-4 acute GVHD. Documented/biopsy proven acute GVHD is graded according to MAGIC grading. Cumulative incidence curves will be used to estimate acute GVHD.
Incidence of severe chronic GVHD | Up to day 180 post-HCT
  Will evaluate sever chronic GVHD. Documented/biopsy proven chronic GVHD is scored according to National Institutes of Health consensus staging. Cumulative incidence curves will be used to estimate chronic GVHD.
NRM | From HCT to death from other causes than disease relapse or progression, assessed up to day 365 post-HCT
  Will evaluate occurrence of NRM. Cumulative incidence curves will be used to estimate NRM.
Relapse | From HCT to the first observation of disease relapse or progression, assessed up to day 365 post-HCT
  Will evaluate time to relapse. NRM is the competing risks event. Cumulative incidence curves will be used to estimate relapse.
Overall survival (OS) | From HCT to the date of death regardless of cause, assessed up to day 365 post-HCT
  Will evaluate OS. OS is censored at the last follow-up if the last known status is alive. Kaplan-Meier curves will be used to estimate OS.
CMV-specific T cell immunity | Up to day 365 post-HCT
  Will evaluate levels and kinetics of CMV-specific T cell immunity, combined with immunophenotyping and functional studies. Repeated measures analysis of variance analyses will be used for immunological functions over time.

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Northside Hospital, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts